CLINICAL TRIAL: NCT04813549
Title: Evaluation of Fibromyalgia Syndrome and Its Effect on Quality of Life in Rheumatoid Arthritis Patients in Our Clinic
Brief Title: Evaluation of Fibromyalgia Syndrome and Its Effect on Quality of Life in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, YILDIZ GONCA DOGRU, RESIDENT OF PHYSICAL MEDICINE AND REHABILITATION, Ahi Evran University Education and Research Hospital
Other Study IDs: 2021-05/50
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis; Fibromyalgia; Fibromyalgia, Secondary
Keywords: fibromyalgia; rheumatoid arthritis; fibromyalgia, secondary
MeSH Terms: conditions — Arthritis, Rheumatoid; Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis patients: Rheumatoid arthritis patients will be evaluated in terms of the presence of secondary fibromyalgia and its effect on the quality of life, at their admission.

SUMMARY:
Rheumatoid arthritis is a chronic, autoimmune, systemic inflammatory disease with a prevalence of approximately 1%. With a lifetime development rate of 3.6%, rheumatoid arthritis is seen 1.7% more in women than in men. Although there are no diagnostic criteria for rheumatoid arthritis, ACR / EULAR 2010 classification criteria are frequently used in diagnosis. Symptom duration, number of swollen joints, acute phase reactants and serology are used in these criteria. Fibromyalgia syndrome is characterized by chronic widespread pain, fatigue, exercise disorders and cognitive impairment. Although the prevalence of fibromyalgia syndrome in the general population is between 2-4%, it is one of the most common conditions encountered by rheumatologists. A treat to target strategy is recommended in rheumatoid arthritis disease management. This approach suggests close monitoring of disease activity and treatment change in cases where the goal is not achieved. The prevalence of fibromyalgia in rheumatoid arthritis patients was found to be 5-52% in meta-analyzes due to the heterogeneity of fibromyalgia criteria used in studies. This study, it was aimed to evaluate the effect of secondary fibromyalgia syndrome, which is frequently found in rheumatoid arthritis and characterized by symptoms such as fatigue and widespread pain, on rheumatoid arthritis disease activation and patients' quality of life.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic, autoimmune, systemic inflammatory disease with a prevalence of approximately 1%. With a lifetime development rate of 3.6%, rheumatoid arthritis is seen 1.7% more in women than in men. Synovial joints are the primary involvement site of the disease, and due to insufficient control of the disease, irreversible joint damage and disability may develop. Although there are no diagnostic criteria for rheumatoid arthritis, ACR / EULAR 2010 classification criteria are frequently used in diagnosis. Symptom duration, number of swollen joints, acute phase reactants and serology are used in these criteria.

Fibromyalgia syndrome is characterized by chronic widespread pain, fatigue, exercise disorders and cognitive impairment. Although the prevalence of fibromyalgia syndrome in the general population is between 2-4%, it is one of the most common conditions encountered by rheumatologists. The prevalence of fibromyalgia increases with age and is more common in women, with a female: the male ratio between 2:1 to 30:1, depending on which diagnostic criteria are applied.

The first approved classification criteria for fibromyalgia syndrome was developed in 1990 by the American College of Rheumatology (ACR). These criteria include chronic widespread pain for more than 3 months and evaluation of 18 sensitive points. Although it was developed for classification, it was also used as a diagnostic criterion by most rheumatologists. Updated diagnostic criteria excluding sensitive point evaluation were published by ACR in 2010. Common pain index and symptom severity score were used in these criteria. In 2011, these criteria were modified with criteria including the physician's assessment of somatic symptoms. The 2010 and 2011 criteria evaluate symptom severity and 'being fibromyalgia' using the common pain index and symptom severity scale.

There are 2 main groups in fibromyalgia, these are; primary fibromyalgia and secondary fibromyalgia due to a comorbid disease. Primary fibromyalgia is more common and characterized by local pain that initially spreads later. Differential diagnosis is difficult in these individuals because of the common symptoms of rheumatological diseases such as pain and fatigue. Centralized pain may develop with inflammatory arthritis or as a result of the disease. Chronic inflammation can mediate central pain from peripheral pain that can cause symptoms in fibromyalgia. In animal models, pro-inflammatory cytokines such as Tumor Necrosis Factor and Interleukin-6 have been associated with abnormal central pain processing and widespread pain sensitivity.

In Rheumatoid Arthritis(RA) patients, the presence of fibromyalgia syndrome was found 2.1 times more frequently in patients who were Rheumatoid Factor negative than those who were positive, and 3.0 times more frequently in patients who were positive in anti-citrullinated protein antibody (ACPA) seronegative. It is thought that in seronegative patients, clinicians may be less likely to diagnose RA or attribute the RA prodroma symptom as fibromyalgia syndrome. Also alternatively, fibromyalgia syndrome may be the underlying diagnosis in some seronegative cases. In another study investigating the presence of secondary fibromyalgia syndrome in patients with early inflammatory arthritis; it was found that ACPA negative patients had fibromyalgia syndrome more frequently than seropositive patients. The authors hypothesized that this might be caused by ACPA-positive patients were treated more aggressively and disease control was reached earlier, or clinicians were more likely to diagnose fibromyalgia in ACPA-negative patients.

A treat to target strategy is recommended in RA disease management. This approach suggests close monitoring of disease activity and treatment change in cases where the goal is not achieved. In randomized studies, with a treat to target strategy, patients have been found to have a decrease in radiological progression, in disease activity, an increase in physical function and quality of life.

The prevalence of fibromyalgia in rheumatoid arthritis patients was found to be 5-52% in meta-analyzes due to the heterogeneity of fibromyalgia criteria used in studies.When the 2010/2011 criterion was used, the prevalence was found to be higher than the 1990 criteria. (24% vs 18%)Despite this heterogeneity, a strong relationship was found between DAS28 and comorbid fibromyalgia. As DAS28, disease activity index such as SDAI( simplified disease activity index) and CDAI (clinical disease activity index) were found to be correlated with comorbid fibromyalgia.

This study, it was aimed to evaluate the effect of secondary fibromyalgia syndrome, which is frequently found in rheumatoid arthritis and characterized by symptoms such as fatigue and widespread pain, on rheumatoid arthritis disease activation and patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with rheumatoid arthritis,
* who can read and write in Turkish,
* participant's admission participating in the study,
* participants who do not have exclusion criteria

Exclusion Criteria:

* participant's refusal to participate in the study,
* lack of cooperation due to cognitive impairment,
* participant's who have a neurological disease,
* presence of drug abuse,
* presence of malignancy in any organ or system,
* serious psychiatric problems (psychosis, etc.),
* the presence of another rheumatological disease other than Rheumatoid Arthritis,
* serious and unstable metabolic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Diagnosis of fibromyalgia syndrome | Participant's admission
  For the diagnosis of fibromyalgia syndrome, "Widespread Pain Index and Symptom Severity Scale", which are the ACR criteria published in 2010, will be used.Widespread Pain Index; The number of painful areas is calculated in the last 1 week. How many areas has the patient had will be calculated. Scoring is between 0-19. Symptom Severity Scale; Scoring is between 0-12. The presence of fatigue, tired awakening, cognitive symptoms, and somatic symptoms will be evaluated by the clinician, and the level of each in the last 1 week will be recorded as (0 = normal, 1 = mild, 2 = moderate, and 3 = severe).
  A patient satisfies diagnostic criteria for fibromyalgia if the following 3 conditions are met:
  1. Widespread Pain Index ≥7 and Symptom Severity Scale ≥5 or Widespread Pain Index 3-6 and Symptom Severity Scale ≥9
  2. Symptoms have been present at a similar level for at least 3 months.
  3. The patient does not have a disorder that would otherwise explain the pain
Evaluation of participant's anxiety and depression | Participant's admission
  Participant's anxiety and depression will be measured with the Hospital Anxiety and Depression Scale (HADS). The Scale contains 14 questions. (7 anxiety and 7 depression) Each question is scored 0 to 3.
  8-10 scores mild, 11-14 scores moderate, 15-21 severe Anxiety and depression score will be measured separately.
Evaluation of participant's quality of life | Participant's admission
  Participant's quality of life will be measured with Short Form-36 Quality of Life Questionnaire
Assessment of the current health status of fibromyalgia syndrome | Participant's admission
  The current health status of fibromyalgia syndrome will be evaluated with Fibromyalgia Impact Questionnaire (FIQ)
Evaluation of rheumatoid arthritis disease activity | Participant's admission
  Rheumatoid arthritis disease activity will be evaluated by DAS28-CRP (C Reactive Protein)
Evaluation of rheumatoid arthritis remission | Participant's admission
  Boolean index criteria will be used for detect the remission.

SECONDARY OUTCOMES:
Evaluation of widespread body pain | Participant's admission
  Widespread body pain will be questioned with Visual Analog Scale. Visual Analog Scale is determined by measuring the distance (mm) on the 10 cm line, between anchor and the patient's mark. Providing a range of scores from 0-100.A higher score indicates greater pain intensity.
  No pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Evaluation of tender points for the presence of pain | Participant's admission
  Tender points are located in clusters on both sides of the body, both above and below the waist. These are in occiput, lower cervical, upper trapezius,supraspinatus muscle, second rib, lateral epicondyle, gluteal region, great trochanter, medial of the knee.

CONTACTS AND LOCATIONS:
Overall Officials: FIGEN TUNCAY, PROF.,M.D., Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kirsehir Ahi Evran University Hospital, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao SS, Duffield SJ, Goodson NJ. The prevalence and impact of comorbid fibromyalgia in inflammatory arthritis. Best Pract Res Clin Rheumatol. 2019 Jun;33(3):101423. doi: 10.1016/j.berh.2019.06.005. Epub 2019 Jul 17. PMID 31703796
- [Background] Gist AC, Guymer EK, Eades LE, Leech M, Littlejohn GO. Fibromyalgia remains a significant burden in rheumatoid arthritis patients in Australia. Int J Rheum Dis. 2018 Mar;21(3):639-646. doi: 10.1111/1756-185X.13055. Epub 2017 Mar 13. PMID 28296177
- [Background] Bas DB, Su J, Wigerblad G, Svensson CI. Pain in rheumatoid arthritis: models and mechanisms. Pain Manag. 2016;6(3):265-84. doi: 10.2217/pmt.16.4. Epub 2016 Apr 18. PMID 27086843